CLINICAL TRIAL: NCT04945421
Title: The Phase Ib/II, Open-label, Multicenter Study of IBI310 (Anti-CTLA4 mAb) in Combination With Sintilimab in Patients With Recurrent/Metastatic Nasopharyngeal Carcinoma That Failed Prior Anti-PD-1/PD-L1 Therapy
Brief Title: IBI310 in Combination With Siltilimab in Subjects With Anti-PD-1/PD-L1 Resistance R/M NPC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI310F201
Record Dates: First submitted 2021-06-07; First posted 2021-06-30 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: NPC
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab and IBI310 (single arm) (Experimental): The test group will be treated with either (IBI310 3 mg/kg IV d1, Q3W combined with sintilimab 100 mg IV d1, Q3W) or( IBI310 1 mg/kg IV d1, Q3W combined with sintilimab 200 mg IV d1, Q3W) for up to 4 cycles, and then sintilimab 200 mg IV d1, Q3W until progressive disease, intolerable toxicity, start of a new antitumor treatment, withdrawal of informed consent, loss to follow-up, death or other situations requiring termination of treatment specified in the protocol, whichever occurs first.
  Interventions: Drug: Sintilimab; Drug: IBI310

INTERVENTIONS:
Drug: Sintilimab — (IBI310 3 mg/kg IV d1, Q3W combined with sintilimab 100 mg IV d1, Q3W) or( IBI310 1 mg/kg IV d1, Q3W combined with sintilimab 200 mg IV d1, Q3W) for up to 4 cycles, and then sintilimab 200 mg IV d1, Q3W until progressive disease, intolerable toxicity, start of a new antitumor treatment, withdrawal of informed consent, loss to follow-up, death or other situations requiring termination of treatment specified in the protocol, whichever occurs first.
Drug: IBI310 — (IBI310 3 mg/kg IV d1, Q3W combined with sintilimab 100 mg IV d1, Q3W) or( IBI310 1 mg/kg IV d1, Q3W combined with sintilimab 200 mg IV d1, Q3W) for up to 4 cycles, and then sintilimab 200 mg IV d1, Q3W until progressive disease, intolerable toxicity, start of a new antitumor treatment, withdrawal of informed consent, loss to follow-up, death or other situations requiring termination of treatment specified in the protocol, whichever occurs first.

SUMMARY:
This is a phase 1b/II, open label, multicenter study of IBI310 (Anti-CTLA4 mAb) in combination with Sintilimab in patients with recurrent/metastatic Nasopharyngeal Carcinoma that failed prior Anti-PD-1/PD-L1 therapy

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years;
2. ECOG 0 ~ 1;
3. Histologically/cytologically confirmed R/M NPC;
4. Failed to prior Anti-PD-1 resistance;
5. Adequate organ and bone marrow function;
6. Expected survival ≥12 weeks;
7. Female subjects of childbearing age or male patients whose sex partners are women of childbearing age should take effective contraceptive measures throughout the treatment period and within 6 months after the last administration;
8. Subjects who sign the written informed consent form, and can abide by the visits and related procedures specified in the protocol.
9. At least 1 measurable lesion according to the Response Evaluation Criteria in Solid Tumors Version 1.1(RECIST V1.1).

Exclusion Criteria:

1. Had tumors other than NPC within the past 5 years.
2. Had allogeneic organ or stem cell transplantation.
3. The presence of uncontrolled life-threatening illness
4. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
5. Patients who have used large doses of glucocorticoids, anti-cancer monoclonal antibodies, and other immunosuppressive agents within 4 weeks.
6. HIV positive.
7. Patients with significantly lower heart, liver, lung, kidney and bone marrow function.
8. Severe, uncontrolled medical conditions and infections.
9. At the same time using other test drugs or in other clinical trials.
10. Refusal or inability to sign informed consent to participate in the trial.
11. Other treatment contraindications.
12. Emotional disturbance or mental illness, no civil capacity or limited capacity for civil conduct.
13. Hepatitis B surface antigen (HBsAg) positive and HBVDNA ≥1000cps/ml.
14. Patients with positive HCV antibody test results can only be included in the study when the polymerase chain reaction of HCV RNA is negative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
ORR(Objective response rate) | Up to 2 years
  Investigator evaluated ORR per RECIST V1.1

SECONDARY OUTCOMES:
DOR(Duration of Response) | Up to 2 years
  defined as the time from the first documented objective response to the first documented progressive disease or death of any cause, whichever occurs first;
PFS (Progress Free Survival) | Up to 2 years
  defined as the time from randomization to the first documented progressive disease or death of any cause, whichever occurs first;
OS (Overall Survival) | Up to 2 years
  defined as the time from randomization to death of any cause in subjects without receiving any immunotherapy outside the study protocol for first-line treatment of advanced HCC;
DCR(Disease control rate) | Up to 2 years
  defined as the proportion of patients whose best response is CR, PR, and stable disease (SD) non-CR/non-PD
TTR(Time to progress) | Up to 2 years
  defined as the time from randomization to the first documented and confirmed objective response (CR or PR)
TEAE(Treatment Emergent Adverse Event)/SAE(Serious Adverse Event) | Up to 2 years
  Incidence and severity of treatment-emergent: which is evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, v5.0, 2017) grade;
Changes of Quality of life, according to EORTC QLQ-C30 | Up to 2 years
  According to EORTC QLQ-C30
Changes of Quality of life, according to EORTC QLQ-H&N35 | Up to 2 years
  According to EORTC QLQ-H&N35
ADAs | Up to 2 years
  The immunogenicity of IBI310 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China